CLINICAL TRIAL: NCT04721600
Title: Evaluation of the Evoke Radiofrequency Device for Improvement of Skin Appearance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: InMode MD Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: DO609576A
Record Dates: First submitted 2020-12-24; First posted 2021-01-22 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2024-06-11 (Actual); Status verified 2024-06

CONDITIONS: Skin Laxity
MeSH Terms: conditions — Cutis Laxa

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- treatment (Experimental): Subjects aged 35-75, healthy adults with visible signs of aging, seeking skin laxity treatments. three treatments
  Interventions: Device: Evoke Radiofrequency Device

INTERVENTIONS:
Device: Evoke Radiofrequency Device — Enrolled subjects will undergo up to 3 successive bi-weekly (every 2 weeks) treatments.Treatment area will include face and under chin

SUMMARY:
Evaluation of the Evoke Radiofrequency Device for Improvement of Skin Appearance

DETAILED DESCRIPTION:
The aim of the study is to evaluate the safety, efficacy, patient comfort, and patient satisfaction after Evoke treatment

ELIGIBILITY:
Inclusion Criteria:

* - Signed informed consent to participate in the study.
* Female and male subjects, 35 and 75 years of age at the time of enrolment
* If female, not pregnant, lactating and must be either post-menopausal, surgically sterilized, or using a medically acceptable form of birth control at least 3 months prior to enrolment (i.e., oral contraceptives, contraceptive implant, barrier methods with spermicide or abstinence).
* In addition, negative urine pregnancy test as tested before each treatment and at the last visit for women with childbearing potential (e.g. not menopause).
* General good health confirmed by medical history and skin examination of the treated area.
* Willing to have photographs and images taken of the treated areas to be used de-identified in evaluations, publications and presentations.
* The patients should be willing to comply with the study procedure and schedule, including the follow up visit, and will refrain from using any other aesthetic treatment methods for the last 6 months and during the entire study period.

Exclusion Criteria:

* - Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body.
* Permanent implant in the treated area such as metal plates and screws, silicone implants or an injected chemical substance, unless deep enough in the periostal plane.
* Current or history of skin cancer, or current condition of any other type of cancer, or premalignant moles.
* Severe concurrent conditions, such as cardiac disorders, epilepsy, uncontrolled hypertension, and liver or kidney diseases.
* Pregnancy and nursing.
* Impaired immune system due to immunosuppressive diseases such as AIDS and HIV, or use of immunosuppressive medications.
* Patients with history of diseases stimulated by heat, such as recurrent Herpes Simplex in the treatment area, may be treated only following a prophylactic regimen.
* Poorly controlled endocrine disorders, such as diabetes or thyroid dysfunction.
* Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.
* History of skin disorders, keloids, abnormal wound healing, as well as very dry and fragile skin.
* History of bleeding coagulopathies or use of anticoagulants in the last 10 days.
* Any surgery in treated area within 3 months prior to treatment.
* Six months delay is required if other recent treatments like light, CO2 laser or RF were performed on the same area.
* Use of Isotretinoin (Accutane®) within 6 months prior to treatment.
* As per the practitioner's discretion, refrain from treating any condition that might make it unsafe for the patient

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2022-07-28 (Actual); Study Completion 2022-07-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Dover, MD, Principal Investigator — Skincare physicians
Locations (1):
- Skincare physicians, Chestnut Hill, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Labadie JG, Chilukuri S, Cohen J, Kilmer S, Lupo M, Rohrich R, Dover JS. Noninvasive Hands-free Bipolar Radiofrequency Facial Remodeling Device for the Improvement of Skin Appearance. Dermatol Surg. 2023 Jan 1;49(1):54-59. doi: 10.1097/DSS.0000000000003666. Epub 2022 Dec 8. PMID 36533797

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment
Started | 15
Completed | 12
Not Completed | 3

BASELINE CHARACTERISTICS:
Population: Subjects aged 35-75, healthy adults with visible signs of aging, seeking skin laxity treatments.
Arm/Group | Treatment
Number analyzed (Participants) | 15
Age, Continuous [Mean (Standard Deviation); unit: years] — Subject age by years
  years | 58 (9.05)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Baseline and 6 Month Face Photographs Correctly Identified by Two Blind Evaluators
Time Frame: 6 months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment
Number analyzed (Participants) | 9
Participants | 7

2. Secondary Outcome: Investigator Assessment of the Skin Appearance
Description: Evaluate Investigator assessment of the skin appearance comparing pre and post-treatment using 0 - 4 -points Likert scale at 6 months follow up visits.
Time Frame: month 6
Population: level of the patients' improvement at 6 months post-treatment. Investigators utilized a scale anchored by 0 (no difference) and 4 (significantly marked improvement).
Measure: Median (Full Range); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 7
units on a scale | 2.4 [0 to 4]

3. Secondary Outcome: Subject Assessment of Change and Satisfaction With the Procedure
Description: patients assessed their satisfaction with the procedure at 6 months post-treatment. Patients utilized a scale anchored by -2 (very disappointed) and 2 (very satisfied).
Time Frame: month 6
Population: patients assessed their satisfaction with the procedure at 6 months post-treatment. Patients utilized a scale anchored by -2 (very disappointed) and 2 (very satisfied).
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Treatment
Number analyzed (Participants) | 12
units on a scale | 0.18 [-2 to 2]

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Treatment
All-Cause Mortality (participants affected / at risk) | 0/15
Serious Adverse Events (participants affected / at risk) | 0/15
Other Adverse Events (participants affected / at risk) | 1/15
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (N=15)
persistent erythema (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-10-21): https://cdn.clinicaltrials.gov/large-docs/00/NCT04721600/Prot_SAP_001.pdf